CLINICAL TRIAL: NCT05478486
Title: A Single Ascending Dose, Phase I Trial to Assess Safety, Tolerability and Pharmacokinetic Profile of MSP008-22 in Patients With Advanced Solid Tumours
Brief Title: Assessment of Safety, Tolerability and PK Profile of MSP008-22 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Godavari Biorefineries Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Clinexel-GBL-002; CTRI/2022/06/043504 (Other: Clinical Trials Registry-India)
Record Dates: First submitted 2022-07-21; First posted 2022-07-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: Single Ascending Dose; First in Man; FIM; SAD; MSP008; Phase 1

STUDY DESIGN:
Intervention Model Description: At least 3 patients will be enrolled at only one dose level and dosed with one only dose of MSP008-22. Each dosed patient will be evaluated for 72.00 hours post-dose for primary and secondary endpoints (i) If there are no AE or abnormal laboratory results experienced by these three patients, the trial will move to the next dose level (next cohort of 3 different patients), (ii) If in a single Cohort, any one patient experiences any Dose Limiting Toxicity, additional 3 patients will be dosed at the same dose level, (iii) If in a single Cohort, more than 33% of the patients experience Dose Limiting Toxicity, the Cohort will be stopped, and further dose escalation will not happen in the study.
Masking Description: It is an open-label clinical trial with a single treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSP008-22 treatment arm (Experimental): Oral Escalating doses of MSP008-22- total five doses, each in form of a single dose oral formulation/tablet.
  Each trial participant will receive only one single oral dose of 05 identified dose levels of MSP008-22. Intra-patient dose escalation will not be carried out
  Interventions: Drug: MSP008-22

INTERVENTIONS:
Drug: MSP008-22 — It is single group assignment interventional model in this clinical trial, consisting of 5 cohorts of 3 patients in each, to be enrolled such that there exists an overall gender balance for the entire trial and to also ensure including minimum five (5) patients of TNBC and minimum five (5) male patients.
  The trial will be initiated with dosing of a cohort of 03 patient with the Safe starting dose for MSP008-22. Dosing of the patients for the next higher dose cohort will initiate only after: (i) All 03 patients have been recruited in the lower dose Cohort and if a repeat Cohort at this dose level is recommended, another 03 patients have been recruited at same dose level (ii) all dosed patients have completed the allocated study cohort duration, (iii) safety and pharmacokinetic results have been reviewed by the Independent Dose Escalation Committee (DEC) and approved for dose escalation to next cohort.

SUMMARY:
This is the 'first-in-human' clinical trial of the Investigational Medicinal Product (IMP), Tablet formulation for Oral dosing of MSP008-22, a molecule (new chemical entity) with anticancer properties.

DETAILED DESCRIPTION:
This Single Ascending Dose (SAD) clinical trial is designed to evaluate the safety and tolerability of single oral ascending doses of the IMP in patients with Stage IV of advanced solid tumours including but not limited to Breast cancer including Triple-negative breast cancer, Ovarian cancer, Prostate cancer, Head and Neck squamous cell cancer).

The trial will also assess the pharmacokinetic (PK) profile of MSP008-22 in humans.

The safety, tolerability and PK data from this trial will determine the safety of MSP008-22 for dosing in humans in further clinical trials.

As MSP008-22 has shown efficacy in in vitro studies against various cancer cell lines and in prostate and breast cancer cell lines in xenograft studies, the first in human trial of MSP008-22 is planned in patients of 'Stage-IV of Advanced Solid Tumours (Breast cancer including Triple-negative breast cancer, Ovarian cancer, Prostate cancer, Head and Neck squamous cell cancer and other advanced solid tumors).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, willing to provide written informed consent and willing to comply to trial requirements, in age range of 18-60 years (both inclusive), with stage IV - metastatic or unresectable Solid tumours (Breast cancer including TNBC, Ovarian cancer, Prostate cancer, Head and Neck squamous cell cancer).
2. Adequate bone marrow function and hepatic & Renal function
3. Has a performance status of 0 to 1 on Eastern cooperative Oncology Group (ECOG) Performance Scale and a Karnofsky Performance Status (KPS) ≥ 70
4. Adequate laboratory parameters for Haemoglobin levels, Absolute Neutrophil Count (ANC), Platelets, AST/SGOT ≤ 2.5 x ULN (≤ 5 x ULN if known liver involvement/ metastases), ALT/SGPT ≤ 2.5 x ULN (≤ 5 x ULN if known liver involvement/ metastases), Total bilirubin ≤ 1.5 x ULN (unless diagnosis of Gilbert's syndrome in which case < 3.0 times ULN), and Serum creatinine ≤ 1.5 x ULN or estimated GFR ≥ 60 mL/min
5. If male, must agree to use contraception and refrain from donating sperm during the treatment period and for ≥120 days after last dose of trial treatment.
6. If female, is not pregnant or breastfeeding, and agrees to use contraception during the treatment period and for ≥120 days after last dose of trial treatment.

Exclusion Criteria:

1. Patients who have been treated with most recent radiotherapy, immunotherapy, chemotherapy or investigational drugs within ≤10 days or 5 half-lives (whichever is shorter) from enrolment (screening), and/or who have any unresolved NCI Common Terminology Criteria of Adverse Events (CTCAE) v5.0 > Grade 1 treatment-related side effect, with the exceptions of alopecia
2. Major surgery (excluding placement of vascular access) ≤21 days from beginning of the study drug or minor surgical procedures ≤7 days.
3. Primary immunodeficiency affecting cellular immunity and active autoimmune disease with the exception of Type I Diabetes Mellitus, hypothyroidism requiring hormone replacement only, an autoimmune dermatologic condition that is managed without systemic therapy, or autoimmune arthritis that is managed without systemic therapy or documented history of autoimmune syndrome or disease.
4. Chronic medical condition that requires chronic steroid therapy or immunosuppressive medication.
5. Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 10 days post dose
  to assess Tolerability of MSP008-22 in Human
Incidence of dose-limiting toxicities (DLTs) | 10 days post-dose
  to assess Safety of MSP008-22 in Human
Incidence of Treatment Emergent adverse events (TEAE); % of patients who experience at least 1 Treatment Emergent Adverse Event (TEAE); % of patients who discontinue due to TEAE(s). | 30 days post-dose
  to assess Safety of MSP008-22 in Human

SECONDARY OUTCOMES:
Plasma Cmax | 72 hours post dose
  (maximum measured concentration of MSP008-22 in plasma)
Plasma AUClast | 72 hours post dose
  (area under the plasma concentration time curve of MSP008-22 from hour 0 to last sample with measurable plasma concentrations)
Plasma AUCinfinity | 72 hours post dose
  (area under the concentration-time curve of MSP008-22 in plasma over the time interval from 0 extrapolated to infinity)
plasma tmax | 72 hours post dose
  (time from dosing to maximum measured concentration of MSP008-22 in plasma)
Plasma t1/2 | 72 hours post dose
  (terminal half-life of MSP008-22 in plasma)
CL/F | 72 hours post dose
  (total clearance of MSP008-22 in plasma after administration estimated using formula)
Vz/F | 72 hours post dose
  (apparent volume of distribution of MSP008-22 during the terminal phase following administration, estimated using formula)
Ae | 72 hours post dose
  (the total amount of MSP008-22 excreted in urine)
Ae %dose | 72 hours post dose
  (the percent of MSP008-22 recovered in urine)
CLr | 72 hours post dose
  (and the apparent renal clearance of MSP008-22)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Arora, MD, Study Director — Clinexel Life Sciences Pvt. Limited
Locations (1):
- Advanced Centre for Treatment, Research and Education in Cancer (ACTREC) of TATA Memorial Centre, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No